CLINICAL TRIAL: NCT00009815
Title: Phase I Study Of Oral Etoposide In Combination With ORZEL (UFT + Leucovorin) For Advanced Non-Hematological Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura A. Pollice, Clinical Research Manager, University of Pittsburgh
Purpose: Treatment
Other Study IDs: 98-013; CDR0000068412 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-990923; NCI-G00-1902
Record Dates: First submitted 2001-02-02; First posted 2004-04-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Etoposide; Leucovorin; Tegafur

INTERVENTIONS:
Drug: etoposide
Drug: leucovorin calcium
Drug: tegafur-uracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of etoposide when combined with fixed- dose fluorouracil-uracil plus leucovorin calcium in patients with advanced solid tumors. II. Determine possible side effects and toxicity of this regimen in these patients.

OUTLINE: This is a dose escalation study of etoposide. Patients receive oral etoposide daily on days 1-10 and oral fluorouracil-uracil plus oral leucovorin calcium twice a day on days 1-21. Treatment repeats every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of etoposide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity. Patients are followed at 2 months and then periodically for survival.

PROJECTED ACCRUAL: Approximately 25-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor for which no curative or effective therapy is available No symptomatic or uncontrolled brain or leptomeningeal metastases CT scan required if clinical suspicion of CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST no greater than 1.5 times ULN No acute hepatitis Renal: Not specified Cardiovascular: No unstable cardiac disease No history of cardiac arrhythmia (treated or untreated) No new onset crescendo or rest angina (stable exertional angina allowed) Pulmonary: Not specified Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception at least 1 week prior to, during, and for at least 2 weeks after study No known hypersensitivity to fluorouracil-uracil or leucovorin calcium No grade 2 or greater nausea/vomiting or diarrhea No significant neurological or psychiatric condition, including psychotic disorders, dementia, or seizures No active serious infection or septicemia No severe gastrointestinal bleeding No other serious illness or significant medical condition that would preclude study No psychological, familial, or sociological condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered No more than 1 prior chemotherapy regimen Prior fluorouracil and taxanes allowed Prior parenteral etoposide allowed Endocrine therapy: No concurrent anti-cancer hormonal agents Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Prior radiotherapy to brain metastases allowed if stable neurological status achieved within 4 weeks of treatment No concurrent radiotherapy except for palliation of bone or brain metastases or pathological fractures of known lytic disease Surgery: Not specified Other: At least 3 weeks since prior investigational drugs and recovered No other concurrent anticancer drugs No other concurrent investigational therapy No concurrent halogenated antiviral agents such as lodenosine, fialuridine, clevudine, emtricitabine, or sorivudine No concurrent antiarrhythmic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P. Belani, MD, Study Chair — University of Pittsburgh